CLINICAL TRIAL: NCT02034214
Title: Economic Opportunity for Zimbabwean Adolescent Orphans
Brief Title: Shaping the Health of Adolescents in Zimbabwe
Acronym: SHAZ!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: UZ-UCSF Collaborative Research Programme (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mi-Suk Kang Dufour, Assistant Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 037044; R01HD045135 (NIH)
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: HIV
Keywords: HIV; adolescents
MeSH Terms: interventions — Reproductive Health Services

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Intervention (Experimental): Life skills education vocational counseling Economic livelihoods reproductive health services social support
  Interventions: Behavioral: Life skills education; Other: Reproductive health services; Behavioral: Economic livelihoods
- Education and health services alone (Active Comparator): Life skills education Reproductive health services
  Interventions: Behavioral: Life skills education; Other: Reproductive health services

INTERVENTIONS:
Behavioral: Life skills education — The life skills curriculum drew upon Stepping Stones and CDC-Zimbabwe Talk Time, developed with input from the target population. It consisted of 14 modules delivered to groups of 25 over 4-6 weeks on: HIV/STI and reproductive health; relationship negotiation; strategies to avoid violence;and identification of safe and risky places in the community. Participants also attended a six-weeks-long home-based care training conducted through Red Cross Zimbabwe, to gain skills on safely caring for people living with HIV.
Other: Reproductive health services — All participants were provided a health screening at every study visit and were treated for treatable STIs and minor ailments. They received condoms, and contraceptive pills or injectable free upon request. Participants who tested positive for HIV were referred to local clinics, where the study team assisted with ART registration including payment for CD4 tests required for enrolment.
Behavioral: Economic livelihoods — The Livelihoods intervention consisted of financial literacy and a choice of vocational training at local training institutes. Courses were 6-months-long, conducted in English, with a practical and a theoretical component. In spite of encouragement to venture outside of accepted gender norms, the most popular courses were hairdressing, garment-making, and receptionist/secretarial and nurse-aid training. Participants who passed developed business plans that were supported with a micro-grant valued at $100US in the form of capital equipment, supplies or additional training.
  Arms: Full Intervention

SUMMARY:
The SHAZ! study was a randomized trial that compared a package of life skills education, reproductive health care services, and economic livelihood development to a control package of life skills education and reproductive health care services alone. SHAZ! enrolled young women 16 to 19 years old who had been orphaned and who were currently out of school and not infected with HIV. Individuals participated in the project for up to two years.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 19 years old
* out of school
* orphaned
* willing to participate in intervention activities
* living in Chitungwiza

Exclusion Criteria:

* HIV infection
* currently pregnant

Ages: 16 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 367 (Actual)
Dates: Start 2006-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Intervention completion | Within 2 years of follow up
  Completion of the intervention activities

SECONDARY OUTCOMES:
Unintended pregnancy | during 2 year follow up
  Urine pregnancy test positive during 2 year follow up period, and pregnancy intendedness on self reported survey
Incident viral infection with HIV or HSV-2 | During 2 years of follow up
  Blood test for HIV and HSV-2 at each 6 month follow up for 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Dunbar, DrPH, MPH, Principal Investigator — Pangea Global AIDS Foundation
Locations (1):
- South Medical, Chitungwiza, Zimbabwe

REFERENCES:
- [Background] Dunbar MS, Maternowska MC, Kang MS, Laver SM, Mudekunye-Mahaka I, Padian NS. Findings from SHAZ!: a feasibility study of a microcredit and life-skills HIV prevention intervention to reduce risk among adolescent female orphans in Zimbabwe. J Prev Interv Community. 2010;38(2):147-61. doi: 10.1080/10852351003640849. PMID 20391061
- [Background] Kang M, Dunbar M, Laver S, Padian N. Maternal versus paternal orphans and HIV/STI risk among adolescent girls in Zimbabwe. AIDS Care. 2008 Feb;20(2):214-7. doi: 10.1080/09540120701534715. PMID 18293132
- [Background] Krishnan S, Dunbar MS, Minnis AM, Medlin CA, Gerdts CE, Padian NS. Poverty, gender inequities, and women's risk of human immunodeficiency virus/AIDS. Ann N Y Acad Sci. 2008;1136:101-10. doi: 10.1196/annals.1425.013. Epub 2007 Oct 22. PMID 17954681
- [Derived] Dunbar MS, Kang Dufour MS, Lambdin B, Mudekunye-Mahaka I, Nhamo D, Padian NS. The SHAZ! project: results from a pilot randomized trial of a structural intervention to prevent HIV among adolescent women in Zimbabwe. PLoS One. 2014 Nov 21;9(11):e113621. doi: 10.1371/journal.pone.0113621. eCollection 2014. PMID 25415455